CLINICAL TRIAL: NCT02502916
Title: Potential Role of the Enteral Feeding Systems on Early Bacterial Gut Colonization of Preterm Infants
Brief Title: Enteral Feeding and Early Gut Colonization of Preterm Infants
Acronym: PRECOL
Status: Completed | Type: Observational
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Juan M. Rodríguez, Professor, Universidad Complutense de Madrid
Other Study IDs: PROBILAC/12O_2
Record Dates: First submitted 2015-07-12; First posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Premature Birth of Newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — meconium, fecal samples mother's milk donor's milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Preterm infant: Preterm infants born from October 2009 to June 2010 at a gestational age of less than 32 weeks or with birth weight of less than 1,200 g

SUMMARY:
The aim of this study is to evaluate the potential role of the enteral feeding systems on the bacterial colonization of premature infants during their NICU admittance and its evolution after 2 years, which is the age when the infant's gut starts to contain an adult-like microbiota.

DETAILED DESCRIPTION:
First spontaneously evacuated meconium and fecal samples were collected by the medical staff of the Hospital weekly from the diapers of the infants during their stay at the Neonatal Intensive Care Unit.

To evaluate the potential role of the enteral feeding systems as a site for colonization by nosocomial bacteria, and, its impact on early gut colonization of preterm neonates, mother's own milk, donor milk and preterm formula samples were obtained after passing through the external part of the enteral feeding tubes and cultured.

Later, when the infants reached 2 years of age, parents were contacted by phone to provide an additional fecal sample if their infants had not taken antibiotics within the previous 2 months.

ELIGIBILITY:
Inclusion Criteria:

* gestational age of less than 32 weeks or with birth weight of less than 1,200 g

Exclusion Criteria:

* any malformation or suffering from any genetic metabolic disorder

Ages: 2 Hours to 8 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants born from October 2009 to June 2010 at the Hospital 12 de Octubre with a gestational age of less than 32 weeks or with birth weight of less than 1,200 g
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of infants sharing bacterial strains with the milk received by each one | two years
  The meconium and fecal samples of the infants have been analysed microbiologically. In parallel, own's mother milk, donor milk and formula milk have been analyzed microbiologically after their pass through the nasogastric feeding tube. The bacterial strains isolated from fecal samples of each infant have been compared with the bacterial strains isolated from the milk that have received each of them.

SECONDARY OUTCOMES:
Number of bacterial strains shared by each infant and the milk received. | two years
  In each infant the number of the same bacterial strains isolated from fecal samples and milk received have been determined.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Rodriguez, PhD, Principal Investigator — Universidad Complutense Madrid

REFERENCES:
- [Derived] Gomez M, Moles L, Melgar A, Ureta N, Bustos G, Fernandez L, Rodriguez JM, Jimenez E. Early Gut Colonization of Preterm Infants: Effect of Enteral Feeding Tubes. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):893-900. doi: 10.1097/MPG.0000000000001104. PMID 26741949